CLINICAL TRIAL: NCT01396304
Title: Restore Calcium Alginate Dressing, Silver vs Aquacel Ag in the Treatment of Critically Colonized Venous Leg Ulcers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Hollister Wound Care LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4835-W
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Venous Ulcer; Infection
Keywords: leg ulcer; infection; closure; wound dressings
MeSH Terms: conditions — Varicose Ulcer; Infections; Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restore Calcium Alginate Dressing Silver (Experimental): Restore Calcium Alginate Dressing Silver under compression wrap
  Interventions: Device: Restore Calcium Alginate Dressing
- Aquacel Ag Wound Dressing (Active Comparator): Aquacel Ag Wound Dressing under compression wrap
  Interventions: Device: AquaCel Ag Wound Dressing

INTERVENTIONS:
Device: Restore Calcium Alginate Dressing — Wound dressing appropriate for venous leg ulcers. Dressing to be changed minimally once per week.
  Arms: Restore Calcium Alginate Dressing Silver
Device: AquaCel Ag Wound Dressing — Wound dressing appropriate for venous leg ulcers. Dressing to be changed minimally once per week.
  Arms: Aquacel Ag Wound Dressing

SUMMARY:
Calcium alginate dressings with silver have been found to be safe and effective for use for leg ulcers. The primary objective is to compare Restore Calcium Alginate Dressing, Silver to AqualCel Ag Dressing on the following parameters: No further progression toward infection (bioburden), ease of application and removal, and percent progression to closure. The secondary objective is to obtain photographic documentation of the leg ulcers during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Is 18 years or older; male or female.
2. Previous diagnosis of venous insufficiency proven by a positive venous duplex with reflux.
3. Has a venous ulcer with a wound area between 5 cm2 - 40 cm2.
4. Has an ankle brachial index (ABI) >0.8.
5. Has a venous ulcer with duration less than 24 months.
6. Has a venous ulcer which is critically colonized (not infected) based on the Lazareth Study Model. Ulcers are considered to be critically colonized if at least three of the five following signs are present:

   Severe spontaneous pain between two dressing changes,Perilesional erythema,Local edema,Malodour,Heavy Exudation
7. Is currently using Profore as their standard of care.
8. Has not received antibiotics for 6 weeks prior to enrollment.

Exclusion Criteria

1. Has an allergy to one of the components of the dressings (calcium alginate, hydrocolloid [carboxymethylceullose], silver).
2. Is currently on antibiotics.
3. Has a negative venous duplex.
4. Is unable to tolerate 4 layer compression.
5. Is unable to continue contact with the investigator for a period of at least two weeks.
6. Is unwilling or unable to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare Restore Calcium Alginate Dressing, Silver to AqualCel Ag Dressing on the following parameters: No further progression toward infection (bioburden), ease of application and removal, and percent progression to closure. | Observations will be collected over 6 weeks for a total of 7 visits

SECONDARY OUTCOMES:
The secondary objective is to obtain photographic documentation of the venous leg ulcers during the course of the study. | Observations will be collected over 6 weeks in a total of 7 visits.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Kaurs, MSHSA MT NMT, Study Director — Hollister Incorporated
Locations (5):
- United States (5):
  - Palms of Pasadena Hospital, St. Petersburg, Florida
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Wound Institute & Research Center, Dunmore, Pennsylvania
  - Lake Washington Vascular Surgeons, Bellevue, Washington